CLINICAL TRIAL: NCT02449083
Title: Cardiac Magnet Resonance Imaging to Evaluate of Dynamic T2 Preparation Puls by Patient With Shunt or Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Magnet Resonance Imaging to Evaluate of Dynamic T2 Preparation Puls by Patients With Shunt or Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Dr. med. Britta Butzbach, Heinrich-Heine University, Duesseldorf
Other Study IDs: 13-007
Record Dates: First submitted 2015-03-19; First posted 2015-05-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Dynamic T2 Preparation
Keywords: MRI; Shunt; COPD; Dynamic T2 Preparation Puls; new sequences; magnet resonance imaging; ventricular septal defect; Atrial septal defect
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Septal Defects, Ventricular; Heart Septal Defects, Atrial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Arm 1: Patients with indication for MRI and coronary angiography
  Interventions: Procedure: MRI; Procedure: coronary angiography
- Arm 2: Patients with atrioseptal or ventriculoseptal Shunt with indication to coronary angiography
  Interventions: Procedure: MRI; Procedure: coronary angiography
- Arm 3: Patients with chronic obstructive pulmonary disease with indication to coronary angiography
  Interventions: Procedure: MRI; Procedure: coronary angiography

INTERVENTIONS:
Procedure: MRI — MRI
Procedure: coronary angiography — coronary angiography

SUMMARY:
There is preliminary evidence that a dynamic T2 Preparations Puls sequence by cardiac magnet resonance imaging can differentiate between oxygenated and deoxygenated blood.

In adult patients with inborn heart defects this has not yet been researched. Therefore,patients with ventriculoperitoneal shunt, septal and atrio-septal shunt should be examined. Also, patients with chronic obstructive pulmonary disease should be examined.

The aim of this study is the validation of a novel magnet resonance sequence in terms of a distinction of oxygenated blood to deoxygenated blood in comparison to invasive method of measuring cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria:

* patients with atrial septal defect (ASD) or ventricular septal defect (VSD) and COPD
* written informed consent

Exclusion Criteria:

* patients with ST-elevation
* contraindication for MRI
* heavy kidney disease
* pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial septal defect (ASD) or ventricular septal defect (VSD) and COPD, who is planned for MRI and angiography
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
ventricular volumetry | baseline
  ventricular volumetry by Cardiac Magnet Resonance Imaging using dynamic T2 Preparation Puls for arithmetical determination of end-systolic volume, end-diastolic volume, ejection fraction, stroke volume and myocardial weight

SECONDARY OUTCOMES:
oxygen partial pressure | baseline
  Determination of oxygen partial pressure (pO2) during angiography
carbon dioxide partial pressure | baseline
  Determination of carbon dioxide partial pressure (pCO2) during angiography
pH-value | baseline
  Determination of pH-value od blood during angiography
Blood gas analysis | baseline
  Determination of base excess of blood during angiography
Blood gas analysis | baseline
  Determination of oxygen partial pressure (pO2), carbon dioxide partial pressure (pCO2), pH-value, base excess
Major adverse cardiac events | 12 month after procedure
  Major adverse cardiac events: death, new indication for angiography, hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Britta Butzbach, MD, Principal Investigator — Heinrich-Heine University, Duesseldorf
Locations (1):
- University Hospital Duesseldorf, Düsseldorf, Germany